CLINICAL TRIAL: NCT04962126
Title: Frontline Treatment of Follicular Lymphoma With AtezolizUmab and Obinutuzumab With and Without RadiOtherapy
Acronym: FLUORO
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Olivia Newton-John Cancer Research Institute (Other)
Collaborators: Roche Products Pty Limited (Unknown); Austin Health (Other Government); Ballarat Health Services (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FLUORO
Record Dates: First submitted 2021-06-29; First posted 2021-07-14 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Follicular Lymphoma
Keywords: Treatment naive advanced disease; anti PD-L1 antibody; anti-CD20 antibody
MeSH Terms: conditions — Lymphoma, Follicular | interventions — obinutuzumab; atezolizumab

STUDY DESIGN:
Intervention Model Description: Single arm phase II study with addition of involved site radiotherapy treatment in participants who achieve only PR/SD at first response assessment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment naive advanced follicular lymphoma (Experimental): All consenting participants will be receive an intravenous infusion of Obinutuzumab (1000mg) + Atezolizumab (1200mg) q3/52 x 6 cycles (plus 1000mg Obinutuzumab on day 8 and 15 of cycle 1). Responding participants (PR or SD) who do not achieve a CR at the end of cycle 2 will receive involved site radiotherapy (4Gy, 2 fractions) between cycle 3 and 4. At the end of cycle 6 and completion of the induction phase, responding participants (CR/PR/SD) will receive maintenance phase Obinutuzumab (1000mg IV) q8/52 for up to 12 cycles.
  Interventions: Drug: Obinutuzumab 25 MG/1 ML Intravenous Solution; Drug: Atezolizumab 1200 MG/40mL Intravenous Solution; Radiation: 4 Gy in 2 fractions

INTERVENTIONS:
Drug: Obinutuzumab 25 MG/1 ML Intravenous Solution — For intravenous infusion during:
  Induction phase: Day 1, 8 and 15 of cycle 1 & Day 1 of cycle 2-6 (q3/52); Maintenance phase: Day 1 of each cycle (q8/52) for up to 12 cycles.
  Other Names: Gazyva
Drug: Atezolizumab 1200 MG/40mL Intravenous Solution — For intravenous infusion during induction phase only day 1 of each cycle q3/52 for up to 6 cycles.
  Other Names: Tecentriq
Radiation: 4 Gy in 2 fractions — Involved site radiotherapy will only be administered to participants to achieve a PR/SD after at restaging after cycle 2, treatment will be between cycle 3 and 4 of induction treatment.

SUMMARY:
This single-arm phase II interventional study aims to assess disease response to, and toxicity of, a combination of obinutuzumab and atezolizumab, with or without radiotherapy, in treatment naive Follicular Lymphoma.

The study will involve an induction phase and a maintenance phase for responding participants, for up to 24 months. Response to treatment will be monitored using medical imaging and clinical assessment.

DETAILED DESCRIPTION:
This is a single-arm phase II study of obinutuzumab, atezolizumab with or without RT in treatment-naïve advanced FL. Participants will initially receive 2 cycles of induction treatment with obinutuzumab and atezolizumab. During cycle 2, participants will undergo disease assessment by PET/CT scan, results of which will determine further induction treatment. Participants in Complete Medical Response (CMR) according to Lugano criteria will receive an additional 4 cycles of induction treatment. Participants who achieve a partial response (PR), stable disease (SD) or deemed to have minor/asymptomatic progressive disease (PD) will also receive 4 further cycles of induction treatment, with the addition of involved-site RT to residual sites of disease (4Gy in 2 fractions), administered between cycle 3 and cycle 4. Participants with symptomatic PD following 2 cycles of induction treatment will not receive any further study treatment. Further treatment will be at the discretion of the treating clinician.

At the end of the induction phase, disease response will again be assessed by PET/CT scan. All participants in CR, PR or SD will move into the maintenance phase of the study and will receive obinutuzumab for 24 months (up to a total of 12 doses). Participants with PD at the end of induction will cease protocol treatment and further treatment will be as per local guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has provided written informed consent
2. Male or female aged ≥ 18 years or older at written informed consent
3. Histologically proven FL grade 1-3A according to the current World Health Organisation classification (2016) including all morphological variants. The B-cell nature of the proliferation must be verified by the positivity with an anti-CD20 antibody
4. No previous chemotherapy, or other investigational drug for this indication apart from focal RT
5. Stage I disease not amenable to single-agent definitive-dose RT, stage II, III or IV (as per Ann Arbor criteria - see appendix 1), suitable for treatment with non-curative intent
6. At least one site of radiographically measurable disease not previously irradiated (at least one bi-dimensionally measurable site of disease: nodal disease >1.5 cm or an extranodal lesion > 1.0 cm in longest perpendicular diameter)
7. Deemed to need treatment by treating Investigator. Reasons for treatment can include, but are not limited to:

   * Any nodal or extranodal tumour mass >7cm AND/OR multiple extranodal disease sites
   * Involvement of at least 3 sites each with diameter >3cm
   * Symptomatic splenic enlargement
   * Organ involvement/compression
   * Ascites or pleural effusion
   * (LDH) elevated
   * Presence of systemic symptoms
   * Disease progression in preceding 3 months
   * Evidence of marrow infiltration with marrow compromise. (e.g. haemoglobin, WBC or platelet count below lower limit of institutional normal range)
8. Adequate bone marrow function within 7 days prior to registration defined as:

   * ANC ≥1.0x109/L
   * WBC ≥2.0x109/L
   * Platelets ≥100x109/L (with no platelet transfusion in the preceding 14 days)
   * Haemoglobin ≥90 g/L (with no red blood cell transfusion in the preceding 14 days) Unless these are attributed to bone marrow infiltration by lymphoma. In cases were one or more results are lower than those specified above due to bone marrow infiltration by FL, patient may be eligible following consultation with the CPI.
9. Adequate organ function within 7 days prior to registration, defined as

   * Total bilirubin ≤1.5 x upper ULN with the exception of patients with known Gilbert's syndrome may be included if their total bilirubin is ≤3.0 x ULN and direct bilirubin ≤1.5 x ULN)
   * AST and(ALT) ≤3 x ULN
   * Adequate renal function with serum creatinine ≤1.5 x ULN or CrCl ≥ 40mL/min (using Cockroft-Gault formula, see Appendix 2)
   * For patients not receiving therapeutic anticoagulation: INR and aPTT ≤ 1.5 x ULN
   * For patients receiving therapeutic anticoagulation: stable anticoagulant regimen
10. ECOG performance status 0-2 (see Appendix 3)
11. Life expectancy greater than 6 months
12. Patients of childbearing potential must adhere to the following:

    * Female patients of childbearing potential must have a negative serum pregnancy test within 7 days prior to registration Note: A woman is considered to be of childbearing potential if she is postmenarchal, has not reached a postmenopausal state (> 12 continuous months of amenorrhea with no identified cause other than menopause), and is not permanently infertile due to surgery (i.e., removal of ovaries, fallopian tubes, and/or uterus) or another cause as determined by the investigator (e.g., Müllerian agenesis). The definition of childbearing potential may be adapted for alignment with local guidelines or regulations.
    * Female patients of childbearing potential must be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the trial through to 18 months after the last dose of treatment. Women must refrain from donating eggs during this same period.

    Note: The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of contraception.
    * Women must not be breastfeeding during study treatment and for 18 months after the last dose of obinutuzumab/study treatment.
    * Male patients must agree to use an adequate method of contraception for the course of the trial through to 18 months after the last dose of treatment. Men must refrain from donating sperm during this same period.
13. Able to comply with the study protocol requirements and follow-up procedures.

Exclusion Criteria:

1. Patient has grade 3B FL, transformed FL or other indolent lymphoma
2. Requirement for urgent treatment due to life-threatening complications of the disease, for example: Compressive symptoms due to disease (which may or may not be bulky), such as superior vena caval obstruction; significant organ involvement causing compromise of organ function (including but not limited to liver/ renal obstruction, actual or impending spinal cord compression, uncontrolled pleural/pericardial effusions), malignant, symptomatic hypercalcaemia
3. Central nervous system, meningeal involvement, cord compression from lymphoma
4. Prior therapy with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways
5. Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF- α agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:

   * Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study after Medical Monitor confirmation has been obtained
   * Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids (≤ 10mg prednisolone for orthostatic hypotension or adrenal insufficiency are eligible for the study
6. Patients with active, known or suspected autoimmune disease, with the following exceptions:

   * Well controlled type I diabetes mellitus
   * Coeliac disease
   * Residual hypothyroidism due to autoimmune condition only requiring hormone replacement
   * Eczema or vitiligo or psoriasis not requiring systemic treatment and rash covering <10% of body surface area
   * Other conditions not expected to recur in the absence of an external trigger
7. Past history of pneumonitis or lung disease including idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organising pneumonia (i.e., bronchiolitis obliterans, cryptogenic organising pneumonia)
8. Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to registration, unstable arrhythmia, or unstable angina
9. Prior organ transplantation or allogeneic bone marrow transplantation
10. Severe active infection with 4 weeks prior to registration , including, but not limited to, hospitalisation for complications of infection
11. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator
12. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
13. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 18months after the last dose of trial treatment, for women and men respectively. Women of childbearing potential must have a negative serum pregnancy test result within 7 days prior to registration.
14. History of HIV (HIV 1/2 antibodies)
15. Active Hepatitis B (Patients with a negative hepatitis B surface antigen (HBsAg) test and a positive total hepatitis B core antibody test (HBcAg) at screening are eligible for the study provided that the screening hepatitis B virus (HBV) DNA test is negative or undetectable). Patients with known hepatitis B on current antiviral therapy are excluded
16. Active Hepatitis C (Patients are eligible with a negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV RNA test at screening. The HCV RNA test will be performed only for patients who have a positive HCV antibody test)
17. Administration of a live, attenuated vaccine within 4 weeks prior to initiation of study treatment or anticipation that such a live attenuated vaccine will be required during the study. Influenza vaccination should be given during influenza season only (example: approximately March to October in the Southern Hemisphere). Patients must not receive live, attenuated influenza vaccine (e.g., FluMist®) within 4 weeks prior registration or at any time during the study treatment or within 5 months after the last dose of protocol treatment. B-cell recovery should be documented prior to administration of live vaccines.
18. Has a known history of active TB (Bacillus Tuberculosis)
19. History of severe allergic anaphylactic reactions to chimeric or humanised antibodies or fusion proteins
20. Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab formulations
21. Major surgical procedure, other than for diagnosis, within 4 weeks prior registration
22. History of malignancy within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate > 90%), such as adequately treated carcinoma in situ of the cervix, non melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-08-17 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Complete metabolic response rate according to Lugano response criteria | At the end of cycle 6 (each cycle in the induction phase is 21 days)
  Complete metabolic response (according to the Lugano response criteria) rate at end of induction (i.e. 6 cycles of obinutuzumab and atezolizumab with or without RT).

SECONDARY OUTCOMES:
Metabolic response rates according to Lugano and RECIL response criteria | After 2 cycles (each cycle in the induction phase is 21 days), at the end of induction phase (6 cycles or 126 days) and at the end of maintenance phase (up to 2 years).
  Response rates (according to Lugano and RECIL response criteria) after two cycles of obinutuzumab and atezolizumab, at end of induction and end of maintenance.
Progression free survival of treated participants | 0-42 months
  PFS
Overall survival of treated participants | 0-42 months
  OS
Quantification of adverse events (according to CTCAEv5.0), including immune-related AEs (irAEs) in treated participants. | 0-27 months
  Number of participants with treatment-related adverse events as assessed using CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Eliza Hawkes, MBBS, Principal Investigator — Austin Health
Locations (3):
- Australia (3):
  - Ballarat Health Service, Ballarat, Victoria
  - Eastern Health, Box Hill, Victoria
  - Austin Health, Heidelberg, Victoria

IPD SHARING:
Plan to Share IPD: No